CLINICAL TRIAL: NCT02364388
Title: IMAging With Opto-acoustics to downgradE BI-RADS claSsificaTion Relative tO Other Diagnostic Methodologies (MAESTRO)
Acronym: MAESTRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seno Medical Instruments Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MAESTRO-01
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: breast imaging diagnosis; breast ultrasound; Imagio; Seno Medical Instruments, Inc.; Seno; opto-acoustics; OA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imagio IUS gray-scale ultrasound (Active Comparator): Imagio gray-scale ultrasound
  Interventions: Device: Imagio IUS; Device: Imagio OA/US
- Imagio OA/US (Other): Imagio OA/US (opto-acoustic+gray-scale ultrasound)
  Interventions: Device: Imagio IUS; Device: Imagio OA/US

INTERVENTIONS:
Device: Imagio IUS — Imagio diagnostic gray-scale ultrasound
  Other Names: gray-scale ultrasound
Device: Imagio OA/US — Diagnostic opto-acoustic +gray-scale ultrasound
  Other Names: Imagio opto-acoustic + gray-scale ultrasound

SUMMARY:
Imagio breast imaging system, is an opto-acoustic (OA) imaging system designed to concurrently collect images in conjunction with diagnostic ultrasound ( co-registered OA and B-mode imaging). This medical device has CE-marking and is approved for use in Europe and other nations.

This is a post-market, non-randomized multi-center surveillance study.

DETAILED DESCRIPTION:
This is a post-market surveillance study that is prospective, controlled, multi-center, to evaluate if Imagio OA can downgrade BI-RADS ( Breast Imaging-Reporting and Data System) classification following CDU (Conventional Diagnostic Ultrasound) for the visualization and characterization of suspicious masses prior to core needle biopsy (CNB) or excision. Investigators will perform CDU to reach a diagnosis and decision to biopsy. Imagio OA will not be used as the reason to perform or to defer a CNB (Core Needle Biopsy) or excision.

ELIGIBILITY:
Inclusion Criteria

* Female
* 18 years of age or older
* Have an undiagnosed suspicious finding which may include more than one solid or complex cystic suspicious mass, classified by CDU as BI-RADS 4a or 4b within 3 weeks of their baseline Imagio Scan

Exclusion Criteria:

* Have a condition or impediment that could interfere with the intended field of view (within one probe length or 4 cm of the mass), (i.e., breast implants within the previous 12 months, or tattoos)
* Pregnant or lactating
* Patient has received chemotherapy for any type of cancer within 90 days from date of screening CDU

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2016-02-15 (Actual); Study Completion 2016-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Rijnstate Hospital, Arnhem
  - Albert Schweitzer Hospital Dordrecht, Dordrecht
  - Zorggroep Twente, Hengelo
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - University Medical Center Utrecht, Utrecht

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective Enrollment from 5 Sites in the Netherlands
Pre-assignment Details: Subjects with BI-RADS 4A or 4B by Conventional Diagnostic Ultrasound
Period: Overall Study
Arm/Group | Imagio OA/US
Started | 217
Biopsied | 209
Excluded | 8
Completed | 209
Not Completed | 8
Not completed — Protocol Violation | 1
Not completed — Technical Failure | 3
Not completed — No OA/US data | 2
Not completed — No Biopsy | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-diagnose (ITD)
Groups:
- MAESTRO: Baseline Breast Imaging Reporting and Data System (BI-RADS) Score of 4a or 4b
Arm/Group | MAESTRO
Number analyzed (Participants) | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 203
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 202
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 209
Number of Masses [Number; unit: Number of masses] — Masses evaluated by site radiologists as either benign, malignant or high-risk (HR). A HR mass is a mass that is not clearly malignant or benign. Population: Masses for participants in the intent-to-diagnose population. Some participants had more than one mass. Masses were grouped according to diagnosis by central independent histopathology review as malignant, benign, or high risk.
  Number of masses
    Benign masses (3 participants had 2 masses): number analyzed (Participants) | 143
    Benign masses (3 participants had 2 masses) | 146
    Malignant masses (3 participants had 2 masses): number analyzed (Participants) | 64
    Malignant masses (3 participants had 2 masses) | 67
    High-risk masses (2 masses, 2 participants): number analyzed (Participants) | 2
    High-risk masses (2 masses, 2 participants) | 2

OUTCOME MEASURES:

1. Primary Outcome: OA/US Specificity (Downgrade (%) for BI-RADS 4A & 4B) of Benign Masses
Description: Outcome is the percentage of benign masses correctly downgraded by (OA/US) ultrasonography from a suspicious abnormality (4A or 4B) to benign or probably benign (BI-RADS 2 or 3). BI-RADS is the Breast Imaging Reporting and Data System established the American College of Radiology. BI-RADS scores range from 0 to 6, with increase in score indicating an increase in the probability of malignancy. A BI-RADS score of 4 or more indicates the need for biopsy. Specificity is reported with a 96% confidence interval using a normal approximation.
Time Frame: CDU images and decision to biopsy to be done at Screening. OA/US imaging to be done within 10 days of Screening. Biopsy to be done within 30 days of Screening.
Population: The intent-to-diagnose population of participants with benign masses. This is the ITD population of masses for specificity.
Measure: Mean (96% Confidence Interval); unit: percentage of masses
Units Other Than Participants: Masses
Groups:
- MAESTRO: Baseline
Arm/Group | MAESTRO
Number analyzed (Participants) | 143
Number analyzed (Masses) | 146
percentage of masses | 41.1 [33.1 to 49.6]

2. Primary Outcome: OA/US Sensitivity (Upgrade (%) for BI-RADS 4A & 4B) of Malignant Masses
Description: Outcome is the percentage of malignant masses correctly identified by (OA/US) ultrasonography as BI-RADS 4a or higher. BI-RADS is the Breast Imaging Reporting and Data System established the American College of Radiology. BI-RADS scores range from 0 to 6, with increase in score indicating an increase in the probability of malignancy. A BI-RADS score of 4 or more indicates the need for biopsy. Sensitivity is reported with a 96% confidence interval using a normal approximation.
Time Frame: as for outcome 1
Population: The intent-to-diagnose population of participants with malignant masses. This is the ITD population of masses for sensitivity.
Measure: Mean (96% Confidence Interval); unit: percentage of masses
Units Other Than Participants: Masses
Arm/Group | MAESTRO
Number analyzed (Participants) | 64
Number analyzed (Masses) | 67
percentage of masses | 95.5 [86.4 to 98.6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Screening Visit through Biopsy. Biopsy was to be done within 30 days of the Screening Visit.
Arm/Group | MAESTRO
All-Cause Mortality (participants affected / at risk) | 0/217
Serious Adverse Events (participants affected / at risk) | 0/217
Other Adverse Events (participants affected / at risk) | 1/217
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAESTRO (N=217)
Post procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication based on the results obtained at the trial site (or a group of sites), including subsets of data, shall not be made before the first multi-center publication.